CLINICAL TRIAL: NCT05888688
Title: The Imaging Assessment of Sarcopenia Across the Heart Failure Spectrum
Brief Title: The Sarcopenia Study
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0916
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure; Sarcopenia; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction; Type 2 Diabetes; Frailty
Keywords: Heart Failure; Sarcopenia; Frailty; Skeletal Muscle; Magnetic Resonance Imaging; 31-Phosphorous magnetic resonance spectroscopy
MeSH Terms: conditions — Heart Failure; Sarcopenia; Diabetes Mellitus, Type 2; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Skeletal muscle biopsy obtained from the thigh.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients with Heart Failure with Preserved Ejection Fraction (HFpEF): Heart Failure (HF) Patients: Stage A/B HFpEF
  1. Established clinical diagnosis of HFpEF (EF>50%)
  2. Clinically stable for ≥ 3 months (no admissions to hospital)
  3. Age ≥65
  4. Willing to provide written consent for participation in the study.
- patients with Heart Failure with Reduced Ejection Fraction (HFrEF): HF Patients: Stage C/D HFpEF and HFrEF
  1. Established clinical diagnosis of HFpEF (EF>50%) OR HFrEF (EF<40%)
  2. Clinically stable for ≥ 3 months (no admissions to hospital)
  3. Age ≥65
  4. Willing to provide written consent for participation in the study.
- Asymptomatic T2D: 1. Male or female, aged ≥18 and ≤75 years.
  2. Diagnosis of stable T2D (determined by i) formal diagnosis in primary care physician case records, ii) a record of diagnostic oral glucose tolerance test OR glycated haemoglobin level ≥6.5%).
- Healthy Volunteers: 1. Age >18
  2. Able to provide written informed consent

SUMMARY:
The goal of this cross-sectional study is to investigate the prevalence of sarcopenia in patients with Heart Failure. The main question it aims to answer is:

Whether there is a difference in the prevalence of sarcopenia across the spectrum of HFpEF (Heart failure with preserved ejection fraction) and HFrEF (heart failure with reduced ejection fraction).

This is an observational study. The participant population involves patients with heart failure with preserved ejection fraction and heart failure with reduced ejection fraction. Healthy volunteers will be recruited as controls in addition to adults with asymptomatic Type 2 Diabetes.

Participants will undergo the following:

1. Skeletal muscle mass, quality and body composition assessments using magnetic resonance imaging (MRI) and bioelectrical impedance analysis (BIA)
2. Skeletal muscle strength assessments (Dynamometer, FysioMeter, handgrip strength)
3. Skeletal muscle energetics assessment (31p-Spectroscopy pre/post-exercise recovery)

Researchers will compare Heart failure groups with healthy controls and adults with asymptomatic type 2 Diabetes to see if there are significant differences in the strength, mass and quality of skeletal muscle.

DETAILED DESCRIPTION:
Heart failure is a complex condition which affects the hearts' ability to pump blood around the body properly. Due to this complexity, it often affects multiple systems in the body and can impact the quality of life. A proportion of heart failure patients also have muscle weakness, where one can feel fatigued, and weak, and may have trouble balancing and standing. To characterise muscle weakness, it is important to look at skeletal muscle mass, strength, and function. The study will focus on the prevalence of reduced muscle strength or function, using a variety of assessments within patients with heart failure. The prevalence of muscle weakness will be investigated by running assessments to look into muscle strength, a series of simple exercise tests will be run of the calf and thigh, in addition to a walking test, a balance test and a standing test to assess whole body performance. To look at the quality of skeletal muscle, a magnetic resonance imaging (MRI) and spectroscopy session will allow us to investigate the quality of the thigh muscle and the energetics in the calf. Finally, a muscle biopsy will be performed to understand differences in muscle tissue in people with different types of heart failure.

Overall, this study will provide us with unique information on skeletal muscle strength, composition and energetics within patients with heart failure, by looking at the main factors which characterise muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

Heart Failure (HF) Patients: Stage A/B HFpEF

1. Established clinical diagnosis of HFpEF (EF>50%)
2. Clinically stable for ≥ 3 months (no admissions to hospital)
3. Age ≥65
4. Willing to provide written consent for participation in the study.

HF Patients: Stage C/D HFpEF and HFrEF

1. Established clinical diagnosis of HFpEF (EF>50%) OR HFrEF (EF<40%)
2. Clinically stable for ≥ 3 months (no admissions to hospital)
3. Age ≥65
4. Willing to provide written consent for participation in the study. Healthy volunteers

1. Age >18 2. Able to provide written informed consent Asymptomatic T2D

1. Male or female, aged ≥18 and ≤75 years.
2. Diagnosis of stable T2D (determined by i) formal diagnosis in primary care physician case records, ii) a record of diagnostic oral glucose tolerance test OR glycated haemoglobin level ≥6.5%).

Exclusion criteria:

Heart failure

1. Absolute contraindication to MRI
2. Inability to walk/undertake the 6-Minute Walk Test (6MWT)
3. Neuromuscular disorders that may impact skeletal muscle assessment, such as motor neurone disease, multiple sclerosis, skeletal muscle myopathies and myositis
4. Regular or intermittent oral corticosteroid use
5. Untreated hyper or hypothyroidism
6. Heart failure-related hospitalisations in the last 3 months

Healthy volunteers

1. Previous or current signs of HF
2. Risk factors for the development of HF, such as hypertension, diabetes Mellitus or coronary artery disease

Asymptomatic Type 2 Diabetes Mellitus (T2D)

1. Angina pectoris or limiting dyspnoea (>NYHA II)
2. Major atherosclerotic disease: Symptomatic CAD, history of MI, previous revascularisation, stroke/transient ischaemic attack or symptomatic peripheral vascular disease.
3. Atrial fibrillation or flutter.
4. Moderate to severe valvular heart disease.
5. History of heart failure or cardiomyopathy.
6. Type 1 diabetes mellitus (T1DM).
7. Low fasting C-peptide levels suggestive of adult-onset T1DM.
8. Stage III-V renal disease (estimated glomerular filtration rate ≤30ml/min/1.73m2).
9. Absolute contraindications to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four groups of subjects will be recruited, subjects with HFpEF, HFrEF, asymptomatic T2D and metabolically healthy non-diabetic controls. The ongoing studies will allow the co-enrolment of participants. They will be recruited to match age, sex and ethnicity as closely as possible to the HF participants.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Volumetric quadriceps skeletal muscle mass (cm^3) | Through study completion, an average of 3 years
  A comparison of volumetric quadriceps skeletal muscle mass (cm3) using MRI between HFpEF and HFrEF patients

SECONDARY OUTCOMES:
HF symptoms and quality of life | Baseline
  Minnesota Living with Heart Failure (MLWHF) questionnaire
Frailty assessment | Baseline
  Edmonton Frail scale
Comparison of Body composition | Baseline
  Bioelectrical impedance analysis (BIA) measure of Appendicular Skeletal muscle (cm^3/height) mass between patient groups
The difference in Muscle fat fraction (percent) | Baseline
  The difference in Muscle fat fraction (%) using MRI (DIXON sequence) of the quadriceps between patient groups
quadriceps Skeletal muscle strength (N) | Baseline
  The difference in quadriceps Skeletal muscle strength (N) between patient groups
Calf plantar flexor strength (N) | Baseline
  The difference in Calf plantar flexor strength (N) (c-station FysioMeter) between patient groups
Handgrip strength (N) | Baseline
  Differences in Handgrip strength (N) (Jamar Dynamometer) between patient groups
A comparison of post-exercise recovery metabolites | Baseline
  A comparison of post-exercise recovery metabolites: Phosphocreatine and inorganic phosphate ratios (PCr/Pi), and Adenosine Triphosphate (ATP) using 31p-Magnetic Resonance Spectroscopy between patient groups
A comparison in distance (metres) walked during 6MWT | Baseline
  A comparison in distance (metres) walked during Six Minute walk test (6MWT) between patient groups
A comparison of daily physical activity | Baseline
  A comparison of daily physical activity behaviours as measured by accelerometry between patient groups
The Short Physical Performance Battery (SPPB) performance | Baseline
  A comparison of lower extremity physical performance following the SPPB test between patient groups
Sarcopenia assessment | Baseline
  SARC-F (Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls) questionnaire

OTHER OUTCOMES:
quadriceps musculoskeletal Biopsy Analysis | Baseline
  RNA sequencing following biopsy acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Gerry McCann, BSc, MB, ChB, MRCP, MD, Principal Investigator — University of Leicester (UoL)
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] Redfield MM, Borlaug BA. Heart Failure With Preserved Ejection Fraction: A Review. JAMA. 2023 Mar 14;329(10):827-838. doi: 10.1001/jama.2023.2020. PMID 36917048
- [Background] Murphy SP, Ibrahim NE, Januzzi JL Jr. Heart Failure With Reduced Ejection Fraction: A Review. JAMA. 2020 Aug 4;324(5):488-504. doi: 10.1001/jama.2020.10262. PMID 32749493
- [Background] Del Buono MG, Arena R, Borlaug BA, Carbone S, Canada JM, Kirkman DL, Garten R, Rodriguez-Miguelez P, Guazzi M, Lavie CJ, Abbate A. Exercise Intolerance in Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 May 7;73(17):2209-2225. doi: 10.1016/j.jacc.2019.01.072. PMID 31047010
- [Background] Pandey A, Shah SJ, Butler J, Kellogg DL Jr, Lewis GD, Forman DE, Mentz RJ, Borlaug BA, Simon MA, Chirinos JA, Fielding RA, Volpi E, Molina AJA, Haykowsky MJ, Sam F, Goodpaster BH, Bertoni AG, Justice JN, White JP, Ding J, Hummel SL, LeBrasseur NK, Taffet GE, Pipinos II, Kitzman D. Exercise Intolerance in Older Adults With Heart Failure With Preserved Ejection Fraction: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 14;78(11):1166-1187. doi: 10.1016/j.jacc.2021.07.014. PMID 34503685
- [Background] Salmon T, Essa H, Tajik B, Isanejad M, Akpan A, Sankaranarayanan R. The Impact of Frailty and Comorbidities on Heart Failure Outcomes. Card Fail Rev. 2022 Mar 21;8:e07. doi: 10.15420/cfr.2021.29. eCollection 2022 Jan. PMID 35399550
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Tucker WJ, Haykowsky MJ, Seo Y, Stehling E, Forman DE. Impaired Exercise Tolerance in Heart Failure: Role of Skeletal Muscle Morphology and Function. Curr Heart Fail Rep. 2018 Dec;15(6):323-331. doi: 10.1007/s11897-018-0408-6. PMID 30178183
- [Result] Uchmanowicz I, Mlynarska A, Lisiak M, Kaluzna-Oleksy M, Wleklik M, Chudiak A, Dudek M, Migaj J, Hinterbuchner L, Gobbens R. Heart Failure and Problems with Frailty Syndrome: Why it is Time to Care About Frailty Syndrome in Heart Failure. Card Fail Rev. 2019 Feb;5(1):37-43. doi: 10.15420/cfr.2018.37.1. PMID 30847244
- [Result] Kitzman DW, Nicklas B, Kraus WE, Lyles MF, Eggebeen J, Morgan TM, Haykowsky M. Skeletal muscle abnormalities and exercise intolerance in older patients with heart failure and preserved ejection fraction. Am J Physiol Heart Circ Physiol. 2014 May;306(9):H1364-70. doi: 10.1152/ajpheart.00004.2014. Epub 2014 Mar 21. PMID 24658015
- [Result] Kirkman DL, Bohmke N, Billingsley HE, Carbone S. Sarcopenic Obesity in Heart Failure With Preserved Ejection Fraction. Front Endocrinol (Lausanne). 2020 Sep 30;11:558271. doi: 10.3389/fendo.2020.558271. eCollection 2020. PMID 33117276
- [Result] Bilak JM, Gulsin GS, McCann GP. Cardiovascular and systemic determinants of exercise capacity in people with type 2 diabetes mellitus. Ther Adv Endocrinol Metab. 2021 Jan 27;12:2042018820980235. doi: 10.1177/2042018820980235. eCollection 2021. PMID 33552463
- [Result] Kinugasa Y, Yamamoto K. The challenge of frailty and sarcopenia in heart failure with preserved ejection fraction. Heart. 2017 Feb;103(3):184-189. doi: 10.1136/heartjnl-2016-309995. Epub 2016 Dec 9. PMID 27940967
- [Result] Pandey A, Parashar A, Kumbhani D, Agarwal S, Garg J, Kitzman D, Levine B, Drazner M, Berry J. Exercise training in patients with heart failure and preserved ejection fraction: meta-analysis of randomized control trials. Circ Heart Fail. 2015 Jan;8(1):33-40. doi: 10.1161/CIRCHEARTFAILURE.114.001615. Epub 2014 Nov 16. PMID 25399909
- [Result] Hamada T, Kubo T, Kawai K, Nakaoka Y, Yabe T, Furuno T, Yamada E, Kitaoka H; Kochi YOSACOI study. Clinical characteristics and frailty status in heart failure with preserved vs. reduced ejection fraction. ESC Heart Fail. 2022 Jun;9(3):1853-1863. doi: 10.1002/ehf2.13885. Epub 2022 Mar 30. PMID 35355441
- [Result] Visser M, Goodpaster BH, Kritchevsky SB, Newman AB, Nevitt M, Rubin SM, Simonsick EM, Harris TB. Muscle mass, muscle strength, and muscle fat infiltration as predictors of incident mobility limitations in well-functioning older persons. J Gerontol A Biol Sci Med Sci. 2005 Mar;60(3):324-33. doi: 10.1093/gerona/60.3.324. PMID 15860469
- [Result] Oba H, Matsui Y, Arai H, Watanabe T, Iida H, Mizuno T, Yamashita S, Ishizuka S, Suzuki Y, Hiraiwa H, Imagama S. Evaluation of muscle quality and quantity for the assessment of sarcopenia using mid-thigh computed tomography: a cohort study. BMC Geriatr. 2021 Apr 13;21(1):239. doi: 10.1186/s12877-021-02187-w. PMID 33849469
- [Result] Chianca V, Albano D, Messina C, Gitto S, Ruffo G, Guarino S, Del Grande F, Sconfienza LM. Sarcopenia: imaging assessment and clinical application. Abdom Radiol (NY). 2022 Sep;47(9):3205-3216. doi: 10.1007/s00261-021-03294-3. Epub 2021 Oct 23. PMID 34687326
- [Result] Weiss K, Schar M, Panjrath GS, Zhang Y, Sharma K, Bottomley PA, Golozar A, Steinberg A, Gerstenblith G, Russell SD, Weiss RG. Fatigability, Exercise Intolerance, and Abnormal Skeletal Muscle Energetics in Heart Failure. Circ Heart Fail. 2017 Jul;10(7):e004129. doi: 10.1161/CIRCHEARTFAILURE.117.004129. PMID 28705910
- [Result] Kitzman DW, Brubaker P, Morgan T, Haykowsky M, Hundley G, Kraus WE, Eggebeen J, Nicklas BJ. Effect of Caloric Restriction or Aerobic Exercise Training on Peak Oxygen Consumption and Quality of Life in Obese Older Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Jan 5;315(1):36-46. doi: 10.1001/jama.2015.17346. PMID 26746456
- [Result] Molina AJ, Bharadwaj MS, Van Horn C, Nicklas BJ, Lyles MF, Eggebeen J, Haykowsky MJ, Brubaker PH, Kitzman DW. Skeletal Muscle Mitochondrial Content, Oxidative Capacity, and Mfn2 Expression Are Reduced in Older Patients With Heart Failure and Preserved Ejection Fraction and Are Related to Exercise Intolerance. JACC Heart Fail. 2016 Aug;4(8):636-45. doi: 10.1016/j.jchf.2016.03.011. Epub 2016 May 11. PMID 27179829
- [Result] O'Neill S, Weeks A, Norgaard JE, Jorgensen MG. Validity and intrarater reliability of a novel device for assessing Plantar flexor strength. PLoS One. 2023 Mar 31;18(3):e0282395. doi: 10.1371/journal.pone.0282395. eCollection 2023. PMID 37000780
- [Result] Brubaker PH, Nicklas BJ, Houston DK, Hundley WG, Chen H, Molina AJA, Lyles WM, Nelson B, Upadhya B, Newland R, Kitzman DW. A Randomized, Controlled Trial of Resistance Training Added to Caloric Restriction Plus Aerobic Exercise Training in Obese Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2023 Feb;16(2):e010161. doi: 10.1161/CIRCHEARTFAILURE.122.010161. Epub 2022 Oct 31. PMID 36314122
- [Result] Konishi M, Kagiyama N, Kamiya K, Saito H, Saito K, Ogasahara Y, Maekawa E, Misumi T, Kitai T, Iwata K, Jujo K, Wada H, Kasai T, Nagamatsu H, Ozawa T, Izawa K, Yamamoto S, Aizawa N, Makino A, Oka K, Momomura SI, Matsue Y. Impact of sarcopenia on prognosis in patients with heart failure with reduced and preserved ejection fraction. Eur J Prev Cardiol. 2021 Aug 9;28(9):1022-1029. doi: 10.1093/eurjpc/zwaa117. PMID 33624112
- [Result] Sugita Y, Ito K, Yoshioka Y, Sakai S. Association of complication of type 2 diabetes mellitus with hemodynamics and exercise capacity in patients with heart failure with preserved ejection fraction: a case-control study in individuals aged 65-80 years. Cardiovasc Diabetol. 2023 Apr 28;22(1):97. doi: 10.1186/s12933-023-01835-2. PMID 37118820